CLINICAL TRIAL: NCT01357265
Title: A Phase II Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface, Antigen, Inactivated, Influenza Vaccine, Formulation 2011/2012, When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of One Dose of an Inactivated Trivalent Sub-unit Influenza Vaccine Administered to Non-elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71_27S; 2010-024400-98 (EudraCT Number)
Record Dates: First submitted 2011-05-05; First posted 2011-05-20 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Influenza
Keywords: Seasonal Influenza; vaccine
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- 1 (Other): No comparator is administered, only one IM single dose of trivalent subunit inactivated influenza vaccine is administered during the vaccination visit
  Interventions: Biological: Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Influenza Vaccine — This phase II is performed as a multicenter study in adult and elderly subjects. Enrolled subjects received one single IM dose of trivalent subunit inactivated flu vaccine during the vaccination visit, according to the study protocol (follow-up period: until day 22) .

SUMMARY:
This study will evaluate safety and immunogenicity of a sub-unit Influenza vaccine when administered to adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy, adult and elderly volunteers over 18 years

Exclusion Criteria:

Individuals with any serious chronic or acute disease or known or suspected impairment of the immune system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the antibody response to each influenza vaccine antigen at 21 days post-immunization in adult and elderly | 22 days including follow-up period
  To evaluate the antibody response to each influenza vaccine antigen, as measured by Single Radial Hemolysis (SRH) and/or HI at 21 days post-immunization in compliance with the requirements of the current EU recommendations for clinical trials related to yearly licensing of influenza vaccines.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via Dei Vestini, Cheiti
  - Dipartimento di Scienze della Salute Università di Genova, Via Pastore, Genova
  - Distretto Sanitario di Base di Fossacesia, Via Polidoro-Vasto, Lanciano
  - ASL Lanciano - Vasto,, Via S. Spaventa, Lanciano
  - Vaccine and Immunotherapy Research Center Department of Infectious and Tropical Diseases San Raffaele Scientific Institute, Via Stamira d'Ancona, Milano
  - Dipartimento di malattie infettive Ospedale San Gerardo, Via Pergolesi 33, Monza